CLINICAL TRIAL: NCT06077812
Title: NYU Langone Health Headache Center Learning Migraine Self-Management Techniques Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-01149
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Migraine
Keywords: Migraine; Self-Management; Headache; Behavioral Intervention
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-Person Migraine Self-Management (Active Comparator)
  Interventions: Behavioral: RELAXaHEAD Smartphone App; Behavioral: In-Person Training
- Remote Migraine Self-Management (Active Comparator)
  Interventions: Behavioral: RELAXaHEAD Smartphone App; Behavioral: Virtual Training

INTERVENTIONS:
Behavioral: RELAXaHEAD Smartphone App — Participants will receive access to the smartphone application RELAXaHEAD, which contains features for migraine self-management including a headache diary.
Behavioral: In-Person Training — Participants will receive in-person training in migraine self-management techniques.
  Arms: In-Person Migraine Self-Management
Behavioral: Virtual Training — Participants will receive virtual training in migraine self-management techniques.
  Arms: Remote Migraine Self-Management

SUMMARY:
The investigators aim to determine the feasibility of a migraine self-management program.

DETAILED DESCRIPTION:
Patients with migraine seen by neurologists/headache specialists within or affiliated with the NYU Langone Health system will be identified via electronic medical record system, or in person. The investigators will randomize 50 participants to an in-person migraine self-management protocol, or a remote migraine self-management protocol. The investigators will examine benefits through follow-up at 2, 4, and 6 month time points.

ELIGIBILITY:
Inclusion Criteria:

* English speaking. (At this time, the validated app is only available in English.)
* 18-65 years of age
* Meets International Classification of Headache Disorder (ICHD)-3 migraine criteria based on a headache specialist or neurologist
* Headaches for ≥1 year
* Has not begun a new migraine preventative medication in the last month
* Agreement to not make any preventive medication changes from the time of trial start until 3 months after beginning the study (Note - Acute medications may be changed if needed. Changes in preventive and acute medication and the time initiated will be recorded to evaluate the potential for medication confounds)
* 4-29 headache days a month (so the study includes those in whom the investigators typically offer preventive treatment [>4 headache days/month] and those with more frequent migraines including chronic migraine [15 days or more/month] but exclude those with continuous headaches)

Exclusion Criteria:

* Diagnosis of Medication Overuse Headache (MOH)
* Patients who have had Cognitive Behavioral Therapy, Biofeedback, or other Relaxation Therapy for migraine in the past year
* Alcohol or other substance abuse as determined by self-report or prior documentation in the medical record
* Current opioid or barbiturate use
* PHQ-8 scores greater than 15, indicating a conservative score of moderately severe depressive symptoms based on the PHQ-9 (in this group, more intense psychological intervention targeted to the depression may be needed, as depression is a significant predictor of migraine chronification and people with migraine and comorbid depression are more likely to be refractory to migraine treatments and to develop medication overuse headache)
* Unable or unwilling to follow a treatment program that relies on written and audio-taped materials
* Coronary heart disease, heart attack, stroke, diabetes mellitus Type 1 or II
* Pregnant (because hormonal fluctuations in pregnancy can affect migraine outcomes)
* Other physical limitations which would prevent participating in the standard protocol of biofeedback being studied

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Number of In-Person Sessions Attended by Participants in the In-Person Migraine Self-Management Arm | Up to Month 2
Number of Days of At-Home Practice | Up to Month 2
Satisfaction Scores | Month 2
  Assessment of satisfaction with the intervention using a Likert scale from 1 to 5 with 1 being strongly disagree, and 5 being strongly agree; the total score is the response; higher scores indicate greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mia T Minen, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to Dr. Mia Minen (Mia.Minen@nyulangone.org). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Dr. Mia Minen (Mia.Minen@nyulangone.org). To gain access, data requestors will need to sign a data access agreement.